CLINICAL TRIAL: NCT02976246
Title: Effect of Vitamin K2 (MK7) on Cardiovascular and Bone Disease in Dialysis Patients: A Prospective, Randomized Placebo-controlled Double Blind Trial
Brief Title: Effect of Vitamin K2 (MK7) on Cardiovascular and Bone Disease in Dialysis Patients
Acronym: RenaKvit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RenaKvit
Record Dates: First submitted 2016-11-03; First posted 2016-11-29 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Vitamin K Supplementation; Endstage Renal Disease; Cardiovascular Disease; Bone Disease
MeSH Terms: conditions — Cardiovascular Diseases; Bone Diseases | interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- RenaKvit-vessel Active (Active Comparator): One tablet of 360 micrograms vitamin K2 given once daily to examine the effect on vascular calcification
  Interventions: Dietary Supplement: Vitamin K2 (MK7)
- RenaKvit-vessel Control (Placebo Comparator): One tablet of non-active drug given once daily
  Interventions: Other: Placebo
- RenaKvit-bone Active (Active Comparator): One tablet of 360 micrograms vitamin K2 given once daily to examine the effect on bone metabolism
  Interventions: Dietary Supplement: Vitamin K2 (MK7)
- RenaKvit-bone control (Placebo Comparator): One tablet of non-active drug given once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin K2 (MK7) — One tablet of vitamin K2 (MK7) 360 micrograms given once daily.
  Other Names: menaquinon 7; MK7
  Arms: RenaKvit-bone Active; RenaKvit-vessel Active
Other: Placebo — One tablet of placebo given once daily.
  Arms: RenaKvit-bone control; RenaKvit-vessel Control

SUMMARY:
Cardiovascular disease (CVD) is the most frequent cause of death in patients (ptt.) with chronic kidney disease (CKD). Compared to the general population death due to CVD is 10-20 times higher in CKD ptt. being treated with hemodialysis. Vascular calcification and hence arterial stiffness is of great importance for the high incidence of CVD.

CKD ptt. in dialysis treatment also have a 3 times higher risk of bone fractures. Both vertebral and other fractures of low energy are associated with a high mortality.

Matrix Gla Protein (MGP) is an important inhibitor of vascular calcification and Osteocalcin (OC) is an important regulator of bone metabolism. The function of both MGP and OC depend on vitamin K.

Vitamin K is supplied with food. The content is low in food recommended to CKD ptt. which is reflected in very low concentrations of vitamin K in their blood samples. A correlation between vitamin K level, incidence of vascular calcification and bone density has been proven; yet there are no trials elucidating the clinical effect of vitamin K on vascular calcification or bone strength.

The investigators will conduct a randomized placebo controlled trial examining the clinical effects of vitamin K2 on vascular calcification and bone mineralization in order to prevent and treat CVD and bone disease in CKD ptt.

Primary study endpoints:

1. Changes in arterial stiffness assessed by pulse wave examination
2. Changes in bone mineral density (BMD) in distal radius assessed by DXA-scans.

Secondary study endpoints:

Changes in coronary artery and valvular calcification assessed by heart-CT-scans, blood pressure, body composition, total and regional BMD, lateral column/aortic calcification score as well as a panel of correlating blood tests.

DETAILED DESCRIPTION:
BACKGROUND

Vascular calcification is a significant problem among patients (ptt.) with chronic kidney disease (CKD) and the prevalence of aortic calcification is twice as high as the general population e.g. Cardiovascular disease (CVD) is the most frequent cause of death in ptt. with CKD. Death due to CVD is 10-20 times higher in CKD ptt. being treated with hemodialysis compared to the background population. Whereas atherosclerosis is a dominating cause of CVD in the general population CKD ptt. tend to develop medial calcification and hence arterial stiffness which is thought to be of great importance in the high incidence of CVD.

CKD ptt. in dialysis treatment also have a 3 times higher risk of bone fractures compared to the general population. Both vertebral and other fractures of low energy are associated with a high mortality in CKD ptt.

The genesis of the arteriosclerosis is still unresolved but seems to be multifactorial. The impaired kidney function itself and the treatment so far both seem to be of importance. The vitamin K-dependent Gla proteins; Matrix Gla Protein (MGP) and Osteocalcin (OC) are described as the most potent inhibitors of vascular calcification and osteoporosis. Until recently CKD ptt. have been treated with vitamin K antagonists which just adds to the focus on vitamin K in this progressive, vascular calcification- and bone demineralization process.

Vitamin K is supplied with food. It consists of several subtypes, e.g. vitamin K1 which is transformed into K2 during digestion. The recommended diet for CKD ptt. is low on vitamin K which is reflected in very low concentrations of vitamin K in blood samples from CKD ptt. in hemodialysis. A supplement of vitamin K1 or K2 will make activation possible for MGP and OC by increasing the concentration of vitamin K2.

A correlation between vitamin K level and incidence of vascular calcification in dialysis ptt. has been proven; yet there are no trials elucidating the clinical effect of vitamin K on vascular calcification in CKD ptt. There are not any trials elucidating the effect of vitamin K on bone strength or number of fractures in dialysis ptt, although a relation between vitamin K and bone mineral density in dialysis ptt. has been shown and a significant increase in age related bone strength was found in a study by introducing a daily supplement of vitamin K.

OBJECTIVE AND HYPOYHESIS

To examine the clinical effect of vitamin K2(MK7) on arterial stiffness assessed by pulse wave examination and bone mineral density assessed by DXA-scans in a group of dialysis ptt. in order to be able to prevent and treat cardiovascular and bone disease in CKD ptt. in the future.

The hypothesis is that a daily supplement of vitamin K2 (MK7) will reduce the calcification process in larger arteries, coronary arteries and -valves and hence reduce the risk of CVD as well as increase the bone mineral density and hence the frequency of bone fractures.

DESIGN

RenaKvit is an investigator initiated, prospective, randomized, double-blinded, placebo controlled intervention trial performed as a nationally, multicenter trial that will run for 2 years. Data will be compiled after 1 and 2 years.

The trial is divided into two sub-studies; RenaKvit-kar (vessel) (n= 48) and RenaKvit-knogle (bone) (n=123), in which the effect of vitamin K2(MK7) on larger arteries, coronary arteries- and valves and the effect on bone with regards to bone mineral density and frequency of fractures are respectively examined.

PATIENTS AND RECRUITMENT

Ptt. will be equally divided by randomization and hence daily be given a tablet of either vitamin K2(MK7) or placebo. According to the criteria of inclusion ptt. will either join the RenaKvit-vessel or the bone group. If criteria are fulfilled ptt. are to join both vessel and bone groups.

Determined by calculation of statistical power, incl. a level of significance of 5%, a standard deviation of 0,95 and strength of 80%, a minimum of 40 ptt (RenaKvit-vessel) and 140 ptt. (RenaKvit-bone) will be included, thus taking potentially drop-outs in account. Both ptt. in hemo- and peritoneal dialysis treatment will be included.

Ptt. will be recruited by the dialysis departments at Zealand University Hospital Roskilde, Holbaek Hospitals, Aarhus University Hospital and Aalborg University Hospital.

There will be no fee for participating ptt.

MEDICINE

Patients are given a daily tablet of either vitamin K 360 micrograms or placebo during a period of 2 x 12 months. Both types of tablets will be of similar look and content, besides vitamin K2.

METHODS

* Pulse Wave examination: Includes both pulse wave analysis and pulse wave velocity measurements. Done by using SphygmoCor©-pulse wave apparatus. Pulse wave examination is used as a measure of the arterial stiffness and is performed after standardized method.
* 24-hour blood pressure and blood pressure measurements: Done by current Danish guidelines (17).
* Coronary artery and -valve calcification: Assessed by CT-scans of the heart using the Agatston Score.
* Bone Mineral Density: Assessed by DEXA-scans.
* Lateral lumbal x- ray and aortic calcification score: A semi-quantitative scoring system used to describe the plaques on the front and the back of the aorta level with each level of the lumbar vertebrae. The method has been found to be predictive of vascular morbidity and mortality.
* Measuring predictors/establishing a biobank: Partly as "routine tests" during dialysis and partly as special kits developed at Vejle Hospital.

STATISTICS

Both groups will have descriptive statistics performed for as well as the presentation of the total population, stratified for gender, age and weight.

Normal-distributed data will be expressed as mean value +/- standard deviation (SD), while other distributed data also will be expressed as median values (interquartile range; interquartile range, IQR). Categorical values will be expressed in numbers and percentages.

Normal-distributed variables will be compared with Student's t-test. Where found appropriate, logarithmic transformation shall be performed. Non-normally distributed variables will be compared with the Mann Whitney U test. Categorical values are to be compared with the Chi Square test.

Changes within the treatment groups over time will be analyzed by paired analysis, and between the treatment groups compared with the non-paired analysis. Forward stepwise multivariate logistic regression analysis is carried out to correct significant confounders of the primary and secondary endpoints.

Analysis of Cox proportional hazards will be performed from time to first clinical event.

P≤0.05 will be considered statistically significant. All results - negative and positive - are expected to be published in peer-review magazines.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Life expectancy > 2 years
* Written consent following oral information
* Permanent treatment with dialysis ≥ 3 months with either peritoneal or hemodialysis

Exclusion Criteria:

* Treatment with vitamin K or vitamin K-antagonist by the beginning of the trial or 1 months within.
* Chronic GI-malabsorption leading to a slower bowel transit (e.g. Celiac disease, Short bowel syndrome).
* Ongoing malignancy (ongoing treatment/clinical controlled visits or diagnosed less than 5 years ago), excl. Non-Melanoma-Skin-Cancer (NMSC).
* Abuse of alcohol or other euphoric drug.
* Women who are pregnant or breast-feeding and women who are in the childbearing age without contraception.
* Total/subtotal parathyroidectomy
* Treatment with recombined PTH.
* Treatment with bisphosphonates or other anti-osteoporotic drugs (Selective Estrogen Reuptake Modulators (SERM), strontium, renalat, denosumab).

Only RenaKvit-kar (vessel):

* Atrial fibrillation/other arrhythmia of significance
* Aortic stenosis of significance
* Agatston score < 100 by heart-CT-scan
* Bilateral upper arm fistula
* Amputation above metatarsal level

Criteria of withdrawal:

* Kidney transplantation
* Starting treatment with vitamin K-antagonists
* Wish to with draw from the participant
* Unacceptable side effect to ingestion of vitamin K or placebo
* Reasonable suspicion of lacking compliance regarding medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
For RenaKvit-vessel: Changes in arterial stiffness assessed by pulse wave examination reflecting vascular calcification (unit: m/s). | 2 years
For RenaKvit-bone: Changes in bone mineral density (BMD) in the distal radial bone (unit T-score). | 2 years

SECONDARY OUTCOMES:
For RenaKvit-vessel: Changes in coronary vascular and -valve calcification assessed by CT-scans of the heart (unit: Agatston-Score). | 2 years
For RenaKvit-vessel: Changes in vascular calcification measured by changes in blood pressure measurements (unit: mmHg). | 2 years
For RenaKvit-bone: Changes in body composition, BMD in the lumbar column, hip and whole body (unit: T-score). | 2 years
For RenaKvit-bone: Changes in abdominal aortic calcification measured by lateral X-ray of lumbar column (unit: abdominal aortic calcification score). | 2 years

OTHER OUTCOMES:
For both RenaKvit-vessel and bone: Changes in specific biochemical markers in blood related to increase in vitamin K-treatment (unit mol/L) | 2 years
  Measuring levels of vitamin K1, vitamin K2, de-/phosphorylated stages of MGP and OC, PIVKA-II, FGF-23, bone specific alkaline phosphatase, CTx-1, P1NP.
For both RenaKvit-vessel and bone: Changes in non-specific biochemical markers in blood related to increase in vitamin K-treatment (unit/L) | 2 years
  Measuring levels of creatinine, urea, ionic calcium, phosphate, 25-OH vitamin D, 1,25-OH2-vitamin D, PTH, sodium, potassium, total CO2, magnesium, HGB, white cells, platelets, ferritin, iron, transferrin, HS CRP, cholesterol, ALT, LDH, alkaline phosphatase, bilirubin, albumin, APTT, haptoglobin, trombingeneration (CAT), F1 + F2.
For both RenaKvit-vessel and bone: Changes in urine production | 2 years
  Monitoring volume, creatinine, urea, protein, albumin.
For both RenaKvit-vessel and bone: Changes in medication | 2 years
  Monitoring phosphate binders, vitamin D analogues, calcimimetics, antihypertensives, cholesterol-lowering drugs.
For both RenaKvit-vessel and bone: monitoring clinical events expected to have relation to trial outcomes. | 2 years
  Monitoring thromboembolic events, bone fractures, parathyroidectomy, death A selection of clinical events will be monitored (occurrence of bone fractures, thromboembolic events, parathyroidectomy as well as changes in medicine consumption during the trial calculated in DDD) and clinical consultations will be held.
  In order to register a potential change during treatment with vitamin K all of the above mentioned are to be performed regularly.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Marckmann, MDS, Study Director — Zealand University Hospital; Ditte Hansen, MDS, Study Director — Herlev Hospital; Marie Frimodt-Moeller, MDS, Study Director — Steno Diabetes Center Copenhagen
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: Undecided